CLINICAL TRIAL: NCT02421120
Title: A Prospective, Multicenter, Open-Label Study to Assess Population Pharmacokinetics and Safety of Intravenous Ceftolozane/Tazobactam in Adult Cystic Fibrosis Patients Admitted With Acute Pulmonary Exacerbation
Brief Title: Population Pharmacokinetics and Safety of Intravenous Ceftolozane/Tazobactam in Adult Cystic Fibrosis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Joseph L. Kuti, PharmD (Other)
Collaborators: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry); Indiana University Health (Other); University of North Carolina (Other); St. Christopher's Hospital for Children (Other)
Responsible Party: Sponsor-Investigator, Joseph L. Kuti, PharmD, Associate Director, Clinical and Economic Studies, Hartford Hospital
Organization: Hartford Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HHC-2015-0107
Record Dates: First submitted 2015-04-13; First posted 2015-04-20 (Estimated); Results first posted 2017-04-13 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Cystic Fibrosis; Cystic Fibrosis Pulmonary Exacerbation; Pseudomonas Aeruginosa Infection
MeSH Terms: conditions — Cystic Fibrosis; Pseudomonas Infections | interventions — ceftolozane, tazobactam drug combination; ceftolozane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ceftolozane/Tazobactam (Experimental): Ceftolozane/Tazobactam 3 grams every 8 hours intravenously for 4-6 doses
  Interventions: Drug: Ceftolozane/Tazobactam

INTERVENTIONS:
Drug: Ceftolozane/Tazobactam — 1 hour intravenous infusion
  Other Names: Zerbaxa; CXA-101

SUMMARY:
There is established evidence that adult patients with Cystic Fibrosis (CF) may have altered antibiotic pharmacokinetics compared with non-CF patients. Ceftolozane/Tazobactam is a newly approved broad spectrum intravenous antibiotic, which has potent in vitro activity against multidrug resistant Pseudomonas aeruginosa, the most common pathogen implicated in CF pulmonary exacerbations. This study will determine the pharmacokinetics and tolerability of ceftolozane/tazobactam in 20 adult CF patients admitted for a pulmonary exacerbation at one of 4 participating hospitals in the US. Patients will remain on standard of care IV antibiotics and receive 4-6 doses of ceftolozane/tazobactam 3 grams every 8 hours. Blood will be sampled after the final dose to determine concentrations and pharmacokinetics of ceftolozane and tazobactam. Safety and tolerability will be assessed throughout the 3 day study.

DETAILED DESCRIPTION:
Participants will receive 4-6 doses of ceftolozane/tazobactam 3 grams every 8 hours, in addition to standard intravenous antibiotic therapy selected by the site. Just prior and then after the final dose, a total of six blood samples will be collected to measure ceftolozane and tazobactam concentrations. Data will be fit to a population pharmacokinetic model. The final model will be utilized in a Monte Carlo simulation to determine the probability of several different dosing regimens retaining concentrations above the minimum inhibitory concentration (MIC) for at least 39% of the dosing interval. These data will be utilized to determine an optimized dosing regimen for adults with CF.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Documented diagnosis of CF
3. Acute pulmonary exacerbation as the primary reason for admission to the hospital with requirement to receive systemic antibiotic treatment
4. If female, subjects must be non-pregnant and non-lactating. Females can be either not of a child-bearing potential or if of a child-bearing potential, on acceptable modes of birth control such as abstinence from sexual intercourse, oral/parenteral contraceptives, or barrier method

Exclusion Criteria:

1. History of any moderate or severe hypersensitivity or allergic reaction to any β-lactam antibiotic (a history of mild rash to a cephalosporin followed by uneventful re-exposure is not a contraindication)
2. Prior (within 24 hours of first dose of study drug) or concomitant receipt of piperacillin/tazobactam or probenecid
3. History of lung transplant
4. Moderate to severe renal dysfunction defined as a creatinine clearance < 50 mL/min (as calculated by the Cockcroft-Gault equation using actual body weight) or requirement for continuous renal replacement therapy or hemodialysis
5. A hemoglobin less than 8 gm/dl at baseline
6. Any rapidly-progressing disease or immediately life-threatening illness (defined as imminent death within 48 hours in the opinion of the investigator)
7. Any condition or circumstance that, in the opinion of the investigator, would compromise the safety of the patient or the quality of study data
8. Planned or prior participation in any other interventional drug study within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph L Kuti, PharmD, Principal Investigator — Hartford Hospital
Locations (4):
- United States (4):
  - Hartford Hospital, Hartford, Connecticut
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Monogue ML, Pettit RS, Muhlebach M, Cies JJ, Nicolau DP, Kuti JL. Population Pharmacokinetics and Safety of Ceftolozane-Tazobactam in Adult Cystic Fibrosis Patients Admitted with Acute Pulmonary Exacerbation. Antimicrob Agents Chemother. 2016 Oct 21;60(11):6578-6584. doi: 10.1128/AAC.01566-16. Print 2016 Nov. PMID 27550351

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ceftolozane/Tazobactam
Started | 21
Completed | 20
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ceftolozane/Tazobactam
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 25.4 [18 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20
Weight [Mean (Standard Deviation); unit: kilograms] | 53.2 (8.2)
Height [Mean (Standard Deviation); unit: centimeters] | 161.8 (8.29)
Creatinine Clearance [Mean (Full Range); unit: milliliters per minute] | 117.7 [62 to 197]

OUTCOME MEASURES:

1. Primary Outcome: Ceftolozane Clearance
Description: This outcome determines the clearance of ceftolozane over the 8 hour dosing interval.
Time Frame: 0, 1-1.08, 1.25-1.5, 2-3, 4-5, and 7-8 hours after start of final dose
Measure: Mean (Standard Deviation); unit: Liters per hour
Arm/Group | Ceftolozane/Tazobactam
Number analyzed (Participants) | 20
Liters per hour | 4.76 (1.13)

2. Primary Outcome: Ceftolozane Volume of Distribution (Central Compartment)
Description: This outcome determines the volume of distribution of ceftolozane over the 8 hour dosing interval.
Time Frame: 0, 1-1.08, 1.25-1.5, 2-3, 4-5, and 7-8 hours after start of final dose
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Ceftolozane/Tazobactam
Number analyzed (Participants) | 20
Liters | 7.51 (2.05)

3. Primary Outcome: Tazobactam Clearance
Description: This outcome determines the clearance of tazobactam over the 8 hour dosing interval.
Time Frame: 0, 1-1.08, 1.25-1.5, 2-3, 4-5, and 7-8 hours after start of final dose
Measure: Mean (Standard Deviation); unit: Liters per hour
Arm/Group | Ceftolozane/Tazobactam
Number analyzed (Participants) | 20
Liters per hour | 20.51 (4.41)

4. Primary Outcome: Tazobactam Volume of Distribution (Central Compartment)
Description: This outcome determines the volume of distribution of tazobactam over the 8 hour dosing interval.
Time Frame: 0, 1-1.08, 1.25-1.5, 2-3, 4-5, and 7-8 hours after start of final dose
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Ceftolozane/Tazobactam
Number analyzed (Participants) | 20
Liters | 7.85 (2.66)

5. Secondary Outcome: Ceftolozane Probability of Target Attainment at 8 mcg/ml
Description: This simulated outcome indicates the likelihood that ceftolozane will retain drug concentrations above the MIC for >/= 60% of the dosing interval at an MIC of 8 mcg/ml when administered as a 3g (2g ceftolozane/1g tazobactam) every 8 hour dose infused over 1 hour. This analysis is conducted via a Monte Carlo simulation using the population pharmacokinetic parameter estimates and dispersion from the 20 participants who contributed pharmacokinetic data to the study.
Time Frame: 24 hours
Population: The results of this analysis are based on 5000 simulated patients with the same pharmacokinetics to the 20 enrolled participants.
Measure: Number; unit: percent of simulated population
Arm/Group | Ceftolozane/Tazobactam
Number analyzed (Participants) | 20
percent of simulated population | 97.1

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the course of the 3 day study.
Description: Laboratory (chemistry, complete blood count, liver function tests, urinalysis) were completed systematically prior to first dose and within 24 hours after completion of the final pharmacokinetic blood sample. All other adverse events collected when reported by the participant or during daily physical examination.
Arm/Group | Ceftolozane/Tazobactam
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 4/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftolozane/Tazobactam (N=21)
Type I Hypersensitivity Reaction (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Chest tightness and tongue swelling after receipt of first dose.
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Hypokalemia (General disorders) | 2 (2)
Liver Function Test Elevation (Hepatobiliary disorders) | 1 (1)
Vaginal Itching (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No